CLINICAL TRIAL: NCT05468957
Title: A Prospective Randomized Study Comparing Time to Ambulation, Time to Hemostasis and Safety Using a Closure Device Alone an in Conjunction With a Potassium Ferrate Pad Following Transfemoral Catheterization
Brief Title: Comparing Perclose to Statseal in Conjunction With Perclose in Femoral 6 French Arteriotomy Closure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Initiating PI left our institution.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Rushi V. Parikh, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-000700
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Arterial Occlusion; Cardiovascular Diseases; Atherosclerosis; Hematoma
MeSH Terms: conditions — Arterial Occlusive Diseases; Cardiovascular Diseases; Atherosclerosis; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Perclose Only (Active Comparator): Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least one minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. Two hours after the patient has had the PercloseTM device deployed the patient will ambulate. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held and the an ambulation trial will be attempted at least 30 minutes after the subsequent trial. This will be continued until the patient has no bleeding at the time of ambulation.
  Interventions: Device: Perclose
- Perclose with Statseal Device (Experimental): Patients will have a PercloseTM device deployed at the arteriotomy. A Statseal disc will applied and manual pressure will be held for at least one minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. Two hours after the patient has had the PercloseTM device deployed the patient will ambulate. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held and the an ambulation trial will be attempted at least 30 minutes after the subsequent trial. This will be continued until the patient has no bleeding at the time of ambulation.
  Interventions: Device: Perclose; Drug: Statseal

INTERVENTIONS:
Device: Perclose — Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least one minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. Two hours after the patient has had the PercloseTM device deployed the patient will ambulate. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held and the an ambulation trial will be attempted at least 30 minutes after the subsequent trial. This will be continued until the patient has no bleeding at the time of ambulation.
  Other Names: Suture based hemostasis device
Drug: Statseal — Patients will have a PercloseTM device deployed at the arteriotomy. A Statseal disc will applied and manual pressure will be held for at least one minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. Two hours after the patient has had the PercloseTM device deployed the patient will ambulate. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held and the an ambulation trial will be attempted at least 30 minutes after the subsequent trial. This will be continued until the patient has no bleeding at the time of ambulation.
  Other Names: potassium ferrate disc with topical hydrophilic polymer
  Arms: Perclose with Statseal Device

SUMMARY:
The purpose of this clinical study is to compare how well two different devices for achieving hemostasis perform in patients undergoing transfemoral procedures with 6 French Access. Both devices are approved by the FDA for this use, and have already been used by clinicians on patients undergoing transfemoral procedures. It is believed that the use of both devices in combination compared to the Perclose alone will shorten the time that it takes to 'seal' the artery, resulting in a shorter period of time that patients would need to lay flat.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing diagnostic angiography or PCI with femoral access who undergo PercloseTM closure.
* Catheterization with a 6Fr system
* Those with a planned radial approach will also be enrolled given the possibility of changing to femoral access in the catheterization lab if radial access is not possible given radial artery spasm, significant patient discomfort with a contraindication to greater levels of sedation, inability to transverse guidewire into the aortic root, inability to engage coronary artery or deliver equipment, or other clinically indicated reason.

Exclusion Criteria:

- Candidates for this study will be excluded if any one of the following criteria is true:

* Use of a hemostasis method or device besides PercloseTM (Perclose may not be used in situations of heavy calcification, presence of dissection, etc).
* Patients undergoing catheterization only from the radial, brachial, ulnar, or distal radial (snuffbox) artery approach.
* Use of an anticoagulant other than unfractionated heparin or bivalirudin.
* Any use of glycoprotein inhibitors or cangrelor.
* Use of sheathless guides.
* Any anticipated need for continued anticoagulation post-catheterization, including extended bivalirudin infusion.
* Any active treatment with oral anticoagulants continued during course of procedure.
* Presence of arteriovenous dialysis fistula in the ipsilateral leg.
* Any physical deformity or trauma / injury of the leg that would prevent proper placement or function of the hemostasis band.
* Inability of the patient to personally consent for the study. (no surrogate consent)
* Cardiogenic shock, emergent procedures (high risk myocardial infarctions), or any clinical instability as assessed by the physician performing the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Time to Ambulation | Within 30 minutes of discharge or 24 hours post procedure (± 1 hour), whichever occurs first.
  From the time of manual compression after PercloseTM deployed until ambulation is initated after hemostasis is achieved.

SECONDARY OUTCOMES:
Time to Discharge | At least 15 minutes after abultation occurs for those in the outpatient setting.
  From the time of manual compression after PercloseTM deployed until discharge order is activated.
Time to hemostasis | Within 30 minutes of discharge or 24 hours post procedure (± 1 hour), whichever occurs first
  From the time of manual compression after PercloseTM deployed until hemostasis is achieved without complication.
Percent of patients with hematoma | Within 30 minutes of discharge or 24 hours post procedure (± 1 hour), whichever occurs first
  Presence of small <5cm, medium 5-10cm, or large >10cm hematoma based on physical exam or diagnostic imaging.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Ronald Reagen, Los Angeles, California
  - UCLA Santa Monica, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided